CLINICAL TRIAL: NCT00929981
Title: Medrol® In Contact Dermatitis: A Prospective Study To Assess The Safety And Effectiveness Of Medrol In Contact Dermatitis In Indian Subjects
Brief Title: A Study To Assess Safety And Effectiveness Of Medrol In Contact Dermatitis In Indian Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0121004
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Results first posted 2011-12-26 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Dermatitis, Contact
Keywords: Contact Dermatitis; Allergic Dermatitis
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oral Methylprednisolone
  Interventions: Drug: Tablet Methylprednisolone (4 or 16 mg)

INTERVENTIONS:
Drug: Tablet Methylprednisolone (4 or 16 mg) — Oral Methylprednisolone tablets (4mg, 16mg) will be given as per locally approved prescribing information

SUMMARY:
This study will be a prospective, non-interventional, single arm and open label study, in patients with contact dermatitis requiring systemic steroid therapy with a purpose to obtain the real life effectiveness and tolerability of Medrol in treating contact dermatitis in Indian patients. Patients with contact dermatitis who have been prescribed for Medrol will be enrolled into the study and will be followed up for the resolution of symptoms

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for enrollment in this study, patients must be prescribed oral Medrol tablets (4mg and 16 mg) for contact dermatitis as per the locally approved prescribing information
* Medrol tablets, will be prescribed to the patient by the physician according to his/her usual practice. The decision to prescribe Medrol tablet will necessarily precede and will be independent of the decision to enroll patient into the study
* Only those patients, who are ready to sign an informed consent, will be included in the study
* Subject can be contacted through telephone

Exclusion Criteria:

* Patients who have any other dermatological or systemic condition that may interfere or confound with the study outcome measurements
* Patients taking any oral steroid preparation or immunomodulators or have taken any such oral medication during last 15 days before enrollment. NSAIDs (Non Steroidal Anti-Inflammatory Agents) are excluded from the list
* Any contraindication to Medrol tablet use. Contraindications of Medrol use are systemic fungal infections and known hypersensitivity to components
* Participation in other studies within last 1 month before the current study begins and/or during study participation
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been prescribed oral Medrol Tablets (4 or 16 mg) for treatment of contact dermatitis will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- India (3):
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Ludhiana, Punjab

RESULTS

PARTICIPANT FLOW:
Groups:
- Medrol: Medrol tablets 4 milligram (mg) and 16 mg were given orally as per locally approved prescribing information. The duration of therapy was flexible.
Period: Overall Study
Arm/Group | Medrol
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Medrol
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Treatment Status (Success/Failure) of Contact Dermatitis (CD) at the Second Follow-up Visit
Description: The signs and symptoms of CD were rated on Physician's Global Assessment (PGA) 5-point scale (range, 0 - 4 scale): 0 - no clinically relevant reaction; 1- macular erythema with induration; 2 - weak (non-vesicular) reaction with erythema, infiltration, and possible papules; 3 - strong (edematous or vesicular) reaction; 4 - extreme (spreading, bullous, ulcerative) reaction. "Success" was defined as a score of 0 or 1 and "failure" was defined as a score of 2, 3, or 4.
Time Frame: Second follow-up visit (Day 5-28)
Population: Full analysis set (FAS) population included all participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Medrol
Number analyzed (Participants) | 80
Percentage of Participants
  Success | 93.8 [86.01 to 97.94]
  Failure | 6.30 [2.06 to 13.99]

2. Secondary Outcome: Treatment Status (Success/Failure) of CD at the First Follow-up Visit
Description: The signs and symptoms of CD were rated on PGA 5-point scale (range, 0 - 4 scale): 0 - no clinically relevant reaction; 1- macular erythema with induration; 2 - weak (non-vesicular) reaction with erythema, infiltration, and possible papules; 3 - strong (edematous or vesicular) reaction; 4 - extreme (spreading, bullous, ulcerative) reaction. "Success" was defined as a score of 0 or 1 and "failure" was defined as a score of 2, 3, or 4.
Time Frame: First follow-up visit (between Day 6 to 10 after start of treatment)
Population: FAS population included all participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Medrol
Number analyzed (Participants) | 80
Percentage of Participants
  Success | 52.50 [41.02 to 63.79]
  Failure | 47.50 [36.21 to 58.98]

3. Secondary Outcome: Treatment Status (Success/Failure) of CD at the Third Follow-up Visit
Description: as for outcome 2
Time Frame: Third follow-up visit (between Day 6 to 10 after EOT)
Population: FAS population included all participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Medrol
Number analyzed (Participants) | 80
Percentage of Participants
  Success | 100.00 [95.49 to 100.00]
  Failure | 0 [0 to 0]

4. Secondary Outcome: Treatment Status (Success/Failure) of CD at the Final Follow-up Visit
Description: as for outcome 2
Time Frame: Final follow-up visit (between Day 25 to 35 after EOT)
Population: FAS population included all participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Medrol
Number analyzed (Participants) | 80
Percentage of Participants
  Success | 100.00 [95.49 to 100.00]
  Failure | 0 [0 to 0]

5. Secondary Outcome: Change From Baseline in Participant-rated Clinical Severity Score of Lesions at First, Second, Third and Final Follow-up Visits
Description: Participant-rated clinical severity score of lesions rated the severity of all symptoms in the past 24 hours on an 11-point Numerical Rating Scale (NRS) where 0 = No lesions and 10 = Most severe possible lesions.
Time Frame: Baseline,First Follow-up(between Day 6-10 of start of treatment),Second(Day 5-28),Third(between Day 6-10 after EOT),Final(between Day 25-35 after EOT)
Population: FAS population included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Medrol
Number analyzed (Participants) | 80
Units on a scale
  Baseline | 6.8 (1.62)
  Change at first follow-up | -4.1 (1.86)
  Change at second follow-up | -6.2 (2.09)
  Change at third follow-up | -6.7 (1.68)
  Change at final follow-up | -6.8 (1.60)

6. Secondary Outcome: Change From Baseline in Participant-rated Pruritus Score at First, Second, Third and Final Follow-up Visits
Description: Participant-rated pruritus score of lesions rated the severity of pruritus suffered in the past 24 hours on an 11-point NRS where 0 = no pruritus and 10 = most severe possible pruritus.
Time Frame: as for outcome 5
Population: FAS population included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Medrol
Number analyzed (Participants) | 80
Units on a scale
  Baseline | 7.3 (1.49)
  Change at first follow-up | -4.2 (2.15)
  Change at second follow-up | -6.3 (2.32)
  Change at third follow-up | -7.1 (1.60)
  Change at final follow-up | -7.2 (1.47)

7. Secondary Outcome: Change From Baseline in Investigator-rated Total Signs and Symptoms of CD Score at First, Second, Third and Final Follow-up Visits
Description: Investigator-rated total signs and symptoms score of CD included pruritus, erythema, induration, vesiculation, edema or other specific sign or symptom rated on a 5 point scale of 0 - 4 (0=none, 1=mild, 2=moderate, 3=severe, 4=extreme) with a total score of 0 - 20 (lower score was preferred).
Time Frame: as for outcome 5
Population: FAS population included all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Medrol
Number analyzed (Participants) | 78
Units on a scale
  Baseline | 9.2 (2.64)
  Change at first follow-up | -5.6 (2.56)
  Change at second follow-up | -8.3 (3.11)
  Change at third follow-up | -9.0 (2.72)
  Change at final follow-up | -9.1 (2.69)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Medrol
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 1/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medrol (N=80)
Dermatitis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.